CLINICAL TRIAL: NCT02540317
Title: Internet-based Cognitive Behavior Therapy for Stress Disorders: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Associate professor, phd, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ICBT for stress
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Adjustment Disorder; Burnout Syndrome
MeSH Terms: conditions — Adjustment Disorders; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment, Internet-based CBT (Experimental): Internet-based treatment with therapist support using an asynchronous messaging system. The treatment is comprised of 12 modules (similar to chapters) and the treatment is 12 weeks long. The treatment is based on cognitive behavior therapy. Participants will be stratified based on diagnosis, i.e. adjustment disorder and burnout.
  Interventions: Behavioral: Internet-based CBT
- Waiting list control (No Intervention): The control condition is a waiting list. Participants in this arm receive no active treatment. After 12 weeks on waiting list, participants are crossed over to treatment.

INTERVENTIONS:
Behavioral: Internet-based CBT — Internet-based treatment with therapist support using an asynchronous messaging system. The treatment is comprised of 12 modules (similar to chapters) and the treatment is 12 weeks long. The treatment is based on cognitive behavior therapy
  Arms: Active treatment, Internet-based CBT

SUMMARY:
Stress disorders in form of adjustment disorder and burnout syndrom are highly prevalent and cause substantial suffering. Prior evidence suggest that these disorders may be effectively treated with cognitive behavior therapy (CBT), but access to psychological treatment is limited. One possible solution is to provide therapy via the Internet, which has been shown to be effective for anxiety disorders and depression. In the present study, we will investigate the efficacy of Internet-based CBT (ICBT) for adjustment disorders and burnout syndrom in a randomized controlled trial (N=100). Participants will be randomized to active treatment (n=50) or a control condition on waiting list.

DETAILED DESCRIPTION:
Stress disorders in form of adjustment disorder and burnout syndrom are highly prevalent and cause substantial suffering. Prior evidence suggest that these disorders may be effectively treated with cognitive behavior therapy (CBT), but access to psychological treatment is limited. One possible solution is to provide therapy via the Internet, which has been shown to be effective for anxiety disorders and depression. Internet-based CBT can be described as online bibliotherapy with therapist support via a secure messaging system. In this study psychologists will deliver the treatment. We will investigate the efficacy of Internet-based CBT (ICBT) for adjustment disorder and burnout syndrom in a randomized controlled trial (N=100). Participants will be randomized to active treatment (n=50) or a control condition on waiting list. We expect that participants who receive ICBT will make superior improvements compared to the control condition on measures of stress, burnout, depressive symptoms, general anxiety and general functioning.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study participants must be between 18 and 65 years of age and suffer from primary stress-related disorders by meeting diagnostic criteria for adjustment disorder or burnout syndrome. Participants must have access to a computer and to the Internet, as well as being able to write and write in Swedish.

Exclusion Criteria:

Exclusion criteria include (a) meeting the criteria for another axis-1 diagnosis that is assessed to be the primary area of difficulty, (b) suffering from substance abuse/dependence in the past 6 months, (c) suffering from current or past psychosis or bipolar disorder, (d) moderate to high suicide risk, (e) initiated or changed pharmachological treatment for depression or anxiety in the past month and (f) other on-going psychological treatment for stress-related difficulties, and (g) not having received CBT for stress-related ill-health in the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Perceived stress scale (PSS) | baseline, weekly during treatment, post-treatment (12 weeks), 6 month follow-up
  Change in PSS at post-treatment and follow-up compared to baseline

SECONDARY OUTCOMES:
Shirlom Melamed Burnout Questionnaire (SMBQ) | baseline, weekly during treatment, post-treatment (12 weeks), 6 month follow-up
  Change in SMBQ at post-treatment and follow-up compared to baseline
Insomnia Severity Index (IS) | baseline, weekly during treatment, post-treatment (12 weeks), 6 month follow-up
  Change in ISI at post-treatment and follow-up compared to baseline
Generalized AnxietyDisorder-7 (GAD-7) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in GAD-7 at post-treatment and follow-up compared to baseline
Physical Health Questionnaire-15 (PHQ-15) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in PHQ-15 at post-treatment and follow-up compared to baseline
Montgomery Åsberg Depression Rating Scale - self-rated (MADRS-S) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in MADRS-S at post-treatment and follow-up compared to baseline
Self-rated health (SRH) | baseline, weekly during treatment, post-treatment (12 weeks), 6 month follow-up
  Change in SRH at post-treatment and follow-up compared to baseline
Work Ability Index (WAI) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in WAI at post-treatment and follow-up compared to baseline
Euroqol 5 dimensions (EQ5D) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in EQ5D at post-treatment and follow-up compared to baseline
Brunnsviken Brief Quality of life inventory (BBQ) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in BBQ at post-treatment and follow-up compared to baseline
World Health Organization Disability Assessment Schedule (WHODAS) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in WHODAS at post-treatment and follow-up compared to baseline.
Alcohol Disorders Identification Test (AUDIT) | Baseline
  This instrument will be used for screening purpose only
Sickness questionnaire state (SQ) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in SQ at post-treatment and follow-up compared to baseline
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in TIC-P at post-treatment and follow-up compared to baseline
Karolinska Sleep Questionnaire (KSQ) | baseline, post-treatment (12 weeks), 6 month follow-up
  Change in KSQ at post-treatment and follow-up compared to baseline
Client Satisfaction Questionnaire (CSQ) | Post-treatment (12 weeks)
  Mean and standard deviations will be presented

OTHER OUTCOMES:
Credibility Scale (C-scale) | Week 2 and week 8
  Measures treatment credibility. Mean scores and standard deviations will be presented
Change in Putative mediators | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12

REFERENCES:
- [Derived] Lindsater E, Axelsson E, Salomonsson S, Santoft F, Ljotsson B, Akerstedt T, Lekander M, Hedman-Lagerlof E. Cost-Effectiveness of Therapist-Guided Internet-Based Cognitive Behavioral Therapy for Stress-Related Disorders: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2019 Sep 13;21(9):e14675. doi: 10.2196/14675. PMID 31586370
- [Derived] Lindsater E, Axelsson E, Salomonsson S, Santoft F, Ejeby K, Ljotsson B, Akerstedt T, Lekander M, Hedman-Lagerlof E. Internet-Based Cognitive Behavioral Therapy for Chronic Stress: A Randomized Controlled Trial. Psychother Psychosom. 2018;87(5):296-305. doi: 10.1159/000490742. Epub 2018 Jul 24. PMID 30041167
- [Derived] Axelsson E, Lindsater E, Ljotsson B, Andersson E, Hedman-Lagerlof E. The 12-item Self-Report World Health Organization Disability Assessment Schedule (WHODAS) 2.0 Administered Via the Internet to Individuals With Anxiety and Stress Disorders: A Psychometric Investigation Based on Data From Two Clinical Trials. JMIR Ment Health. 2017 Dec 8;4(4):e58. doi: 10.2196/mental.7497. PMID 29222080